CLINICAL TRIAL: NCT05517837
Title: A Phase 1, Randomized, Multi-Part, First-in-Human Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single and Multiple Doses of BMS-986421 in Healthy Participants
Brief Title: A Phase 1, First-in-Human Study of BMS-986421 in Healthy Participants
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Adverse change in the risk/benefit.
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: IM052-004
Record Dates: First submitted 2022-08-24; First posted 2022-08-26 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Healthy Participants
Keywords: BMS-986421; Safety; Tolerability; Dose Escalation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BMS-986421 Under Fasted Conditions (Experimental)
  Interventions: Drug: BMS-986421
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: BMS-986421 — Specified dose on specified days
  Arms: BMS-986421 Under Fasted Conditions
Other: Placebo — Specified dose on specified days
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the safety and tolerability of BMS-986421 in healthy adult participants.

ELIGIBILITY:
Inclusion Criteria:

* Participants are required to remain in the clinical facility from Day -1 (Part 1) or Day -2 (Part 2) until clinic discharge.
* A negative test for COVID-19, which will be performed in the manner mandated by the clinical site where this study is being conducted, at screening and admission.
* All female participants, Women of Childbearing Potential (WOCBP) and women not of childbearing potential, must have a negative highly sensitive serum pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin (HCG)) at screening and on Day -1 (or Day -2 for Part 2).

Exclusion Criteria:

* Participant was exposed to an investigational drug (new chemical entity) within 30 days preceding the first dose administration, or 5 half-lives of that investigational drug, if known (whichever is longer).
* Vaccination or plans for vaccination with non-live vaccines within 30 days before Day -1 (for Day -2 for Part 2) until the follow-up phone call.
* Donation of blood or blood transfusion within 8 weeks of first study intervention administration.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2022-09-13 (Actual); Primary Completion 2023-07-14 (Actual); Study Completion 2023-07-14 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) | Up to 8 Weeks
Number of participants with physical examination abnormalities | Up to 8 Weeks
Number of participants with vital sign abnormalities | Up to 8 Weeks
Number of participants with electrocardiogram (ECG) abnormalities | Up to 8 Weeks
Number of participants with clinical laboratory abnormalities | Up to 8 Weeks

SECONDARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | Up to 192 hours after each dose
Area under the plasma concentration-time curve from time zero to time last quantifiable concentration (AUC[0-T]) | Up to 192 hours after each dose
Time of maximum observed plasma concentration (Tmax) | Up to 192 hours after each dose

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution - 0001, Cypress, California, United States

IPD SHARING:
Plan to Share IPD: No
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myers Squibb's data sharing policy and process can be found at: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosurecommitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/us/en/home.html